CLINICAL TRIAL: NCT05543486
Title: Clinical Evaluation of the Levitation Knee Brace in Patients With Knee Osteoarthritis: A Pilot Study
Brief Title: Clinical Evaluation of the Levitation Knee Brace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Bone and Joint Health Strategic Clinical Network (BJH SCN) (Unknown); McCaig Institiute of Bone and Joint Health (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Strategy for Patient Oriented Research Support Unit (AbSPORU) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB20-1106
Record Dates: First submitted 2022-09-06; First posted 2022-09-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Brace; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, parallel arm
Who Masked: Outcomes Assessor
Masking Description: Outcomes are assessed by a blinded examiner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Levitation 2 Tri-Compartment Offloader (TCO) knee brace (Experimental): Participants in this group are sized and fitted for a Levitation 2 TCO brace and instructed to wear the brace on their affected limb for a total of 3 or more hours per day for 3 months.
  Interventions: Device: Levitation 2 Tri-Compartment Offloader (TCO) knee brace
- Knee sleeve (Active Comparator): Participants are provided with a off-the-shelf knee sleeve and instructed to wear the sleeve on their affected limb for a total of 3 or more hours per day for 3 months.
  Interventions: Device: Knee sleeve
- Standard of Care Self-Management (No Intervention): Control group practicing conservative self-management of knee osteoarthritis without using a knee device (e.g., hard brace or sleeve) for 3 months.

INTERVENTIONS:
Device: Levitation 2 Tri-Compartment Offloader (TCO) knee brace — Spring Loaded Technology Levitation 2 Tri-Compartment Offloader (TCO) brace containing proprietary spring technology providing a knee extension assist.
  Arms: Levitation 2 Tri-Compartment Offloader (TCO) knee brace
Device: Knee sleeve — Neenca soft knee sleeve comprised of elastic air knit fabric with a silicone padded patella inset and flexible stays on the medial and lateral sides.
  Arms: Knee sleeve

SUMMARY:
Osteoarthritis (OA) is a debilitating disease affecting approximately 1/3 of Canadians over the age of 25. Knee OA typically involves at least 2 of 3 compartments in the knee joint. Conservative treatments include knee braces to manage symptoms and improve joint function. Most knee OA braces are designed to offload one knee compartment, but are not usually indicated for multicompartment knee OA. The Levitation Tri-compartment Offloader (TCO) knee brace stores energy during flexion and provides extension assistance to offload all 3 knee compartments. While there is strong preliminary evidence that the TCO can provide pain relief and improved knee function to users, it is critical to determine whether this brace will have similar benefits for patients with multicompartment knee OA. This pilot randomized control trial evaluates the clinical outcomes of using the TCO in comparison to the current conservative standard of care for knee OA patients.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a debilitating musculoskeletal disease affecting approximately 1/3 of Canadians over age 25. The disease is characterized by loss of cartilage in the afflicted joint and can be a major source of pain, disability, and reduced quality of life. The direct cost of OA in Canada was $2.9 billion CAD in 2010 and is expected to rise to $7.6 billion CAD by 2031. Total knee replacement (TKR) is often used to restore mobility, and the risk for expensive and invasive revision surgery is 2-5 times higher in OA patients younger than 65 years. Thus, finding an alternate early treatment intervention is imperative for societal and economic health. It is well established that excess joint loading is associated with symptoms of knee pain. Existing knee OA (KOA) braces are designed to unload part of the joint to help reduce symptoms of pain and enable patients to participate in physical activity. However, because the majority of KOA braces are designed to offload only one tibiofemoral compartment, they are not indicated for most patients who suffer from patellofemoral (PF) or multi-compartment KOA. The Levitation "Tri-Compartment Offloader" (TCO) knee brace developed by Spring Loaded Technology (SLT) was designed to reduce KOA pain by decreasing compressive forces in all three compartments of the knee with a silicone "liquid spring" providing knee extension assist. The design is predicted to lower the tensile forces of the quadriceps pulling on the knee, thereby decreasing internal joint forces in all three knee compartments. Survey evidence suggests the TCO provides pain relief and improved function to long-term wearers with KOA, especially those with involvement of the PF compartment. However, the generalizability of these benefits to a larger group needs to be investigated through a controlled clinical study involving patients with PF or multi-compartment KOA. The TCO brace provides both a proprioceptive effect as well as a mechanical effect. Soft-shell neoprene knee braces (or 'sleeves') have been shown to reduce pain in KOA patients, believed to be a result of improved proprioception. In order to better isolate and understand the mechanical effect of the extension assist mechanism of the TCO brace on patient outcomes, we require an intervention group with a proprioception intervention only, such as a neoprene sleeve, to remove the potentially confounding effect of proprioception on measured outcomes. Preliminary clinical trial priorities, design and outcome measures have been developed based on clinical outcomes of interest relating to KOA. Participation from key stakeholders including patients, healthcare providers, healthcare administrators and brace manufacturers is critical to ensure research priorities and outcomes are relevant and meaningful. This study represents an opportunity to work directly with patients in the research process, and to evaluate the outcomes of adopting a patient-oriented research approach. Therefore, the focus of this project is to (1) strengthen our preliminary clinical trial plan by refining the priorities, design and desired outcomes, and (2) complete and evaluate a pilot clinical trial based on patient and knowledge-user participation in all phases of the project.

The overall research goal is to conduct a clinical evaluation of the TCO knee brace for treating PF or multi-compartment KOA while incorporating patient participation for optimized study design, implementation and analysis of key outcome measures. This goal will be accomplished across 3 objectives (OB) that coincide with 3 distinct project phases, whereby each project phase is dependent on the outcomes of the previous project phases.

Phase 1 (OB1): Review and improve clinical trial objectives, design and methodology.

Phase 2 (OB2): Perform a pilot trial to evaluate the TCO knee brace in 30 study participants.

Phase 3 (OB3): Interpret study results and create a knowledge translation (KT) plan.

A fourth study objective (OB4) is to evaluate the impact of patient and researcher engagement on the study. This objective will be addressed throughout the duration of the study.

Study Milestones (Specific Aims - SA relating to Objectives).

SA1.1 Recruit patient partners to form the Patient Advisory Committee (PAC).

SA1.2 Plan and conduct a focus group to review clinical trial design and methodology.

SA1.3 Summarize and incorporate patient and researcher feedback into the clinical trial design.

SA2.1 Recruit pilot study participants and assign into an intervention group.

SA2.2 Collect baseline data and 3-month intervention data.

SA2.3 Perform statistical data analysis.

SA3.1 Plan and conduct a focus group to review study results and solicit ideas for dissemination.

SA3.2 Incorporate feedback into interpretation of pilot trial results.

SA3.3 Create and implement knowledge dissemination plan.

SA4.1 Create framework to evaluate patient and researcher engagement.

SA4.2 Implement evaluation tool to evaluate patient and researcher engagement.

SA4.3 Analyze and summarize results of engagement evaluation.

KOA affects over 14 million individuals in North America. In Canada, the economic burden of OA cost the healthcare system approximately $27.5B in 2010. A significant portion of the economic burden is related to indirect costs from loss of employment, tax dollars, and disability compensation. This is largely driven by a lack of appropriate solutions for KOA patients to maintain independence and mobility. The Levitation TCO knee brace represents a promising new technology for reducing pain and maintaining mobility in patients who have, or are developing KOA. Generating scientific evidence on the effectiveness of the TCO brace will allow patients and healthcare providers to make informed decisions regarding their treatment options for KOA. Involving patients directly in the study design, conduct, interpretation and dissemination activities will increase the relevance and utility of results and the overall impact. If proven effective, this solution will allow patients to continue working and living the lifestyle they enjoy for much longer than they would otherwise. Given the high prevalence of KOA, the TCO brace has the potential to significantly improve quality of life for millions of Canadians, while significantly reducing the economic burden of KOA in Canada and beyond.

ELIGIBILITY:
Inclusion Criteria:

* Patellofemoral of combined patellofemoral and tibiofemoral knee osteoarthritis
* Kellgren-Lawrence grade ≥ 2 osteoarthritis (moderate-severe) on weight bearing tunnel view x-ray + skyline
* Experience knee pain that worsens (VAS pain score ≥ 4) with activities such as squatting, rising from seated, and going up and down stairs
* Experience less pain (VAS pain score) in the contralateral knee than in the affected knee during weight-bearing activities
* < 7 degrees of varus/valgus knee alignment
* Knee flexion/extension range of motion from 5-100 degrees minimum
* Between the ages of 18-80
* Able to hear and understand study information and instructions in English
* Must be able to be fit with a Levitation knee brace

Exclusion Criteria:

* History of arthroplasty or high tibial osteotomy in the affected limb
* Surgery (excluding arthroscopy) on either lower limb within last 6 months
* Arthroscopic debridement of the affected knee within last 3 months
* Received corticosteroid injections in last 3 months
* Received hyaluronic acid or platelet-rich plasma (PRP) injections in last 6 months
* History of rheumatoid arthritis
* Symptomatic disease of the hip, ankle, or foot
* History of traumatic onset of knee pain
* A major lower limb injury within the past year requiring physiotherapy or surgery
* Previous fracture of the tibia or femur of the affected limb
* History of diabetic neuropathy or peripheral vascular disease
* Parkinson's or neurodegenerative order that may affect balance / ability to ambulate
* Use of a non-study provided knee brace on the affected limb over the study period
* Known allergy or adverse skin reaction to neoprene
* Open skin wounds present on the leg of the affected side
* Unable to physically or mentally comply with the wearing of a knee brace
* Any contraindications for knee bracing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
VAS pain score - chair rise (3 month) | Change from baseline to 3-month follow up
  Change in VAS pain score from baseline to follow up at 3 months (primary end point).
  Self-reported knee pain intensity experienced over the last week during rising from a seated position, measured using a 0-100 mm visual analogue scale (VAS), where 0 mm represents no pain and 100 mm represents the worst pain imaginable.

SECONDARY OUTCOMES:
VAS pain score - squatting | Change from baseline to 6-week and 3-month follow ups
  Change in VAS pain score from baseline to follow ups at 6 weeks and 3 months.
  Self-reported knee pain intensity experienced over the last week during squatting, measured using a 0-100 mm visual analogue scale (VAS), where 0 mm represents no pain and 100 mm represents the worst pain imaginable.
VAS pain score - stairs | Change from baseline to 6-week and 3-month follow ups
  Change in VAS pain score from baseline to follow ups at 6 weeks and 3 months.
  Self-reported knee pain intensity experienced over the last week during stairs, measured using a 0-100 mm visual analogue scale (VAS), where 0 mm represents no pain and 100 mm represents the worst pain imaginable.
VAS pain score - walking on incline | Change from baseline to 6-week and 3-month follow ups
  Change in VAS pain score from baseline to follow ups at 6 weeks and 3 months.
  Self-reported knee pain intensity experienced over the last week during walking on an incline, measured using a 0-100 mm visual analogue scale (VAS), where 0 mm represents no pain and 100 mm represents the worst pain imaginable.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Change from baseline to 6-week and 3-month follow ups
  Change in KOOS from baseline to follow ups at 6 weeks and 3 months.
  Knee Injury and Osteoarthritis Outcome Score (KOOS) encompasses 42-tiems (question) across 5 sub-scales: Pain (9 items); Symptoms (7 items); Activities of Daily Living Function (17 items); Sport and Recreation Function (5 items); Quality of Life (4 items). Each item uses a Likert scale with five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems). Each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems.
EQ-5D Health-related quality of life score | Change from baseline to 6-week and 3-month follow ups
  Change in EQ-5D health-related quality of life score from baseline to follow ups at 6 weeks and 3 months.
  Health related quality of life score is collected using the 5-item descriptive system of the EQ-5D questionnaire covering five dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems (1), slight problems (2), moderate problems (3), severe problems (4) and extreme problems (5). The level (score) for the five dimensions is combined into a 5-digit number that describes the patient's health state.
30 second chair stand test | Change from baseline to 3-month follow up
  Change in 30 second chair stand test score from baseline to follow up at 3 months.
  The maximum number of sit to stand repetitions from a stationary chair (seat height = 44 cm) that can be completed in 30 seconds.
40m fast-paced walk test | Change from baseline to 3-month follow up
  Change in 40m fast-paced walk test score from baseline to follow up at 3 months.
  The amount of time in seconds it taken to walk a 40 meters along a 10 meter long gait platform, moving as quickly as without running.
Stair climb test | Change from baseline to 3-month follow up
  Change in stair climb test score from baseline to follow up at 3 months.
  The amount of time in seconds to ascend and immediately descend a 5-step staircase (step height = 19 cm) as quickly as possible without running or skipping steps.
Timed up and go test | Change from baseline to 3-month follow up
  Change in stair climb test score from baseline to follow up at 3 months.
  The amount of time in seconds taken to rise from a stationary chair, walk 3 meters forward, turn, walk 3 meters back to the chair, and sit back down in the chair, moving as quickly as possible without running.
6 minute walk test | Change from baseline to 3-month follow up
  Change in 6 minute walk test score from baseline to follow up at 3 months.
  The maximum amount of distance in meters that can be walked in 6 minutes along a 10 meter gait platform, moving as quickly as possible without running.
Quadriceps strength | Change from baseline to 3-month follow up
  Change in quadriceps strength from baseline to follow up at 3 months.
  Quadriceps strength refers to maximal voluntary isometric contraction the quadriceps muscles at 45 degrees of knee bend measured in Newton meters (Nm) using a Biodex Medical Systems dynamometer. Quadriceps strength score is recorded as average peak torque in Nm across 3 maximal quadriceps contractions lasting 3 seconds with a 1 minute rest between contractions.
Hamstrings strength | Change from baseline to 3-month follow up
  Change in hamstrings strength from baseline to follow up at 3 months.
  Hamstrings strength refers to the maximal voluntary isometric contraction of the hamstrings muscles at 15 degrees of knee bend measured as peak torque in Newton meters (Nm) using a Biodex Medical Systems dynamometer. Hamstrings strength score is recorded as average peak torque in Nm across 3 maximal hamstrings contractions lasting 3 seconds with a 1 minute rest between contractions.
EQ-VAS | Change from baseline to 6-week and 3-month follow ups
  Change in EQ-VAS score from baseline to follow ups at 6 weeks and 3 months.
  The EQ VAS records self-rated health on a 0-100 vertical visual analogue scale (VAS), where 0 is labelled as "The worst health you can imagine" and 100 is labelled as "The best health you can imagine."
VAS pain score - chair rise (6 week) | Change from baseline to 6-week follow up
  Change in VAS pain score from baseline to follow up at 6 weeks.
  Self-reported knee pain intensity experienced over the last week during rising from a seated position, measured using a 0-100 mm visual analogue scale (VAS), where 0 mm represents no pain and 100 mm represents the worst pain imaginable.

OTHER OUTCOMES:
Lower Extremity Activity Scale (LEAS) score | Change from baseline to 6-week and 3-month follow ups
  Change in LEAS score from baseline to follow ups at 6 weeks and 3 months.
  Self-reported regular daily activity level, measured using the Lower Extremity Activity Scale (LEAS). The LEAS is a single item questionnaire containing 18 response options that is scored on scale ranging from 1 (confined to bed all day) to 18 (daily vigorous physical activity).
Pre-intervention expectation | Baseline
  Pre-intervention expectation at baseline.
  Pre-intervention expectation for pain relief conferred by the study intervention, measured using a 1-item subset of the Knee Scoring System (KSS) questionnaire with scored on a 5-point Likert scale ranging from 1 (no, not at all) to 5 (yes, a lot).
VAS pain score - associated pain | Change from baseline to 6-week and 3-month follow ups
  Change in VAS pain score of bodily regions with associated pain from baseline to follow ups at 6 weeks and 3 months.
  Self-reported pain intensity over the past week in regions of the body that participants' believe to be related to their knee pain. Response options include the contralateral knee, ipsilateral hip, contralateral hip, ipsilateral ankle, and contralateral ankle. Participants may select "other" to report up to 4 other bodily regions with associated pain, specifying the region. Pain intensity is measured using a 0-100 mm visual analogue scale (VAS), where 0 mm represents no pain and 100 mm represents the worst pain imaginable.
OPUS-CSD | 6-weeks, 3-months
  OPUS-CSD at 6 weeks and 3 months of participants randomized to knee sleeve and Levitation TCO knee brace groups.
  Self-reported satisfaction with knee intervention device measured by the Orthotics Prosthetics User Survey -- Satisfaction with Devices (OPUS-CSD) questionnaire, administered only to participants in the brace or sleeve intervention groups
Device usage | 6-weeks, 3-months
  Device usage time at 6-weeks and 3-months of participants randomized to knee sleeve and Levitation TCO knee brace groups.
  Self-reported average amount of daily knee device usage over the past week in hours and minutes of participants in the brace or sleeve intervention groups.
Medication usage | Change from baseline to 6-week and 3-month follow ups.
  Change in medication usage from baseline to follow ups at 6-weeks 3-months.
  Self-reported medication usage, including average weekly frequency (times per week) and amount (number of pills) of analgesics, non-steroidal anti-inflammatory drugs, topical analgesics, opioid analgesics used in the previous month.
Surgical self-prognosis | Change from baseline to 6-week and 3-month follow ups
  Change in surgical self-prognosis from baseline to follow ups at 6-weeks and 3-months.
  Participants' perceived need to undergo knee replacement therapy in the next 24 months and current plans for knee replacement therapy
Post-intervention expectation | 6-week, 3-months
  Post-intevention expectation at 6 weeks and 3 months.
  Reassessment of pre-intervention expectation for pain relief conferred by the study intervention, measured using a 1-item subset of the Knee Scoring System (KSS) questionnaire with scored on a 5-point Likert scale ranging from 1 (too high- "I'm a lot worse than what I thought") to 5 (too low- "I'm a lot better than I thought").

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Ronsky, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birtwhistle R, Morkem R, Peat G, Williamson T, Green ME, Khan S, Jordan KP. Prevalence and management of osteoarthritis in primary care: an epidemiologic cohort study from the Canadian Primary Care Sentinel Surveillance Network. CMAJ Open. 2015 Jul 17;3(3):E270-5. doi: 10.9778/cmajo.20150018. eCollection 2015 Jul-Sep. PMID 26442224
- [Background] Sharif B, Kopec J, Bansback N, Rahman MM, Flanagan WM, Wong H, Fines P, Anis A. Projecting the direct cost burden of osteoarthritis in Canada using a microsimulation model. Osteoarthritis Cartilage. 2015 Oct;23(10):1654-63. doi: 10.1016/j.joca.2015.05.029. Epub 2015 Jun 5. PMID 26050868
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Felson DT. The sources of pain in knee osteoarthritis. Curr Opin Rheumatol. 2005 Sep;17(5):624-8. doi: 10.1097/01.bor.0000172800.49120.97. PMID 16093843
- [Background] Heekin RD, Fokin AA. Incidence of bicompartmental osteoarthritis in patients undergoing total and unicompartmental knee arthroplasty: is the time ripe for a less radical treatment? J Knee Surg. 2014 Feb;27(1):77-81. doi: 10.1055/s-0033-1349401. Epub 2013 Jul 19. PMID 23873317
- [Background] Budarick AR, MacKeil BE, Fitzgerald S, Cowper-Smith CD. Design Evaluation of a Novel Multicompartment Unloader Knee Brace. J Biomech Eng. 2020 Jan 1;142(1):014502. doi: 10.1115/1.4044818. PMID 31523751
- [Background] Kirkley A, Webster-Bogaert S, Litchfield R, Amendola A, MacDonald S, McCalden R, Fowler P. The effect of bracing on varus gonarthrosis. J Bone Joint Surg Am. 1999 Apr;81(4):539-48. doi: 10.2106/00004623-199904000-00012. PMID 10225800
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant changes in patient reported outcomes in knee and hip osteoarthritis: the minimal clinically important improvement. Ann Rheum Dis. 2005 Jan;64(1):29-33. doi: 10.1136/ard.2004.022905. Epub 2004 Jun 18. PMID 15208174
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Murphy L, Schwartz TA, Helmick CG, Renner JB, Tudor G, Koch G, Dragomir A, Kalsbeek WD, Luta G, Jordan JM. Lifetime risk of symptomatic knee osteoarthritis. Arthritis Rheum. 2008 Sep 15;59(9):1207-13. doi: 10.1002/art.24021. PMID 18759314
- [Background] Suri P, Morgenroth DC, Hunter DJ. Epidemiology of osteoarthritis and associated comorbidities. PM R. 2012 May;4(5 Suppl):S10-9. doi: 10.1016/j.pmrj.2012.01.007. PMID 22632687
- [Background] Cherian JJ, Bhave A, Kapadia BH, Starr R, McElroy MJ, Mont MA. Strength and Functional Improvement Using Pneumatic Brace with Extension Assist for End-Stage Knee Osteoarthritis: A Prospective, Randomized trial. J Arthroplasty. 2015 May;30(5):747-53. doi: 10.1016/j.arth.2014.11.036. Epub 2014 Nov 29. PMID 25499679
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Deshpande BR, Katz JN, Solomon DH, Yelin EH, Hunter DJ, Messier SP, Suter LG, Losina E. Number of Persons With Symptomatic Knee Osteoarthritis in the US: Impact of Race and Ethnicity, Age, Sex, and Obesity. Arthritis Care Res (Hoboken). 2016 Dec;68(12):1743-1750. doi: 10.1002/acr.22897. Epub 2016 Nov 3. PMID 27014966
- [Background] Bombardier C, Hawker GA, Mosher D. The impact of arthritis in Canada: Today and over the next 30 years. Arthritis Alliance of Canda, 2011. https://www.arthritisalliance.ca/images/PDF/eng/Initiatives/20111022_2200_impact_of_arthritis.pdf
- [Background] McGibbon CA, Mohamed A. Knee load reduction from an energy storing mechanical brace: a simulation study. 20th Biennial meeting, Canadian Society of Biomechanics, Halifax, Canada, Aug 2018.
- [Derived] Bishop EL, Bonhomme J, Joffe M, Cowper-Smith C, Ronsky JL, Clark ML. A feasibility randomised trial evaluating the levitation tri-compartment offloader knee brace for multicompartment knee osteoarthritis. Pilot Feasibility Stud. 2025 Jun 13;11(1):81. doi: 10.1186/s40814-025-01660-2. PMID 40514746